CLINICAL TRIAL: NCT00335920
Title: A Prospective, Randomized, Double Blind, Placebo Controlled, Multicenter Study on the Safety and Efficacy of Continuous Infusion of Corticosteroid Delivered Via Catheter in Patients With Idiopathic Sudden Sensorineural Hearing Loss
Brief Title: Safety and Efficacy of Intratympanic Application of Dexamethasone Via Catheter in Patients With Sudden Hearing Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Dr. Dr. h.c. mult. Hans-Peter Zenner, University of Tuebingen, D/o Otorhinolarymgology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOCAL DEX-ISSNHL; Inner ear topical dexamethason
Record Dates: First submitted 2006-06-09; First posted 2006-06-12 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-02

CONDITIONS: Sudden Deafness
Keywords: Sudden Hearing Loss; intratympanic; steroids
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Dexamethasone-dihydrogenphosphate (4mg/ml)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of an intratympanic continuous two-week application of dexamethasone compared to placebo using a temporarily implanted catheter in patients with severe to profound sudden sensorineural hearing loss and insufficient recovery after initial systemic prednisolone therapy.

DETAILED DESCRIPTION:
Patients suffering from unilateral severe to profound sudden sensorineural hearing loss (ISSNHL) or anacusis with no or insufficient recovery after 12-21 days after onset will be treated for 14 days with Dexamethasone or placebo delivered intratympanically via a micro-catheter temporarily implanted into the round window niche and an external mini-pump.

Due to the relatively unknown risks of intratympanic treatment by catheter implantation, a significant spontaneous recovery rate and an existing standard therapy for ISSNHL in Germany (systemic glucocorticoids), patients will only be enrolled into the study if no or insufficient recovery of hearing threshold could be observed after initial systemic therapy.

The study will be carried out until 10 patients per group have been randomized regardless in which study center they have been randomized. After the last patient of these 10 patients per group has reached the endpoint an interim analysis will be done. The statistical estimation of the total number of subjects to be randomized will be completed after this interim analysis by the responsible statistician.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Age is greater than 18 years old and less than 75 years old.
* Diagnosis of unilateral Idiopathic sudden sensorineural hearing loss (i.e. sudden sensorineural hearing loss of unknown etiology
* Sensorineural hearing loss is at least 50 dB or more for three or more frequencies in standard pure tone, bone-conducted audiogram within the range of 500 Hz to 4000 Hz (500, 1000, 2000, 3000 and 4000), 60 dB or more for two of these frequencies or 70 dB or more for any frequency within this range, or a decrease in the SRT to 70 dB or greater (not accounted for by conductive hearing loss) or a drop in speech discrimination score to less than or equal to 30%
* hearing loss occurred within 72 hours
* Hearing loss occurred at least 12 days ago but less than or equal to 21 days ago
* Insufficient recovery of the ISSNHL at least 12 days after onset whether or not the patient received Local Standard Therapy (i.e. Hearing in the contralateral ear is at least 20 dB better than the affected ear in at least three frequencies (any three of 500, 1000, 2000, 3000, 4000 Hz))

Exclusion Criteria:

* Age is less than 18 or greater than 75 years old
* Hearing loss occurred less than 12 days or more than 21 days ago
* Positive pregnancy test, risk of pregnancy (insufficient protection or lactation
* Middle ear inflammation or effusion
* Ear canal inflammation
* Conductive hearing loss of greater than 10 dB
* Sudden bilateral hearing loss
* Presence of any conditions or symptoms which indicate that the hearing loss is not ISSNHL, for example, acoustic trauma, Meniere's disease, fluctuating hearing loss, endolymphatic hydrops, suspected retro-cochlear lesion, hearing loss due to ear surgery, perilymph fistula or barotrauma.
* Pulse synchronic tinnitus (potentially due to glomus jugulare tumor)
* Previous otologic surgery (excluding ventilation tubes)
* History in the past 6 months of ototoxic treatment such as chemotherapy, use of loop diuretics, high dose aspirin, etc.
* Known hypersensitivity, allergy or intolerance to the study medication or any history of severe abnormal drug reaction
* Use of non-permitted treatment during the study
* Intake of experimental drugs or participation in a clinical study within the last 30 days
* Only hearing ear
* History of drug abuse or alcoholism
* History of an ischemic disorder (previous strokes, previous heart attacks, peripheral arterial occlusion disease)
* Patient is not capable of understanding the informed consent form (whether due to its language or for other reasons)
* Any psychiatric syndrome requiring treatment with neuroleptics, antidepressants, hypnotics or anxiolytics which has/have been prescribed within three month preceding inclusion into the study and/or cannot be continued at the same dose during the study
* Any severe (systemic) neurological disease (e.g. Epilepsy, Parkinson's disease, Dementia/Alzheimer's disease, Multiple sclerosis)
* Any reason, in the investigator's opinion, that prohibits inclusion into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pure tone audiometric threshold

SECONDARY OUTCOMES:
Word recognition (speech audiometry)
tinnitus improvement
adverse events (worsening of hearing and/or vertigo and/or tinnitus, middle ear inflammation, pain)

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Zenner, M.D., Principal Investigator — Department of Otorhinolaryngology, University of Tubingen; Stefan K Plontke, M.D., Study Director — Department of Otorhinolaryngology, University of Tubingen
Locations (3):
- Germany (3):
  - St. Vincentius Kliniken, Klinik für HNO Heilkunde, Karlsruhe
  - Department of Otorhinolaryngology, University of Tubingen, Tübingen
  - Bundeswehrkrankenhaus Ulm, Ulm

REFERENCES:
- [Derived] Plontke SK, Lowenheim H, Mertens J, Engel C, Meisner C, Weidner A, Zimmermann R, Preyer S, Koitschev A, Zenner HP. Randomized, double blind, placebo controlled trial on the safety and efficacy of continuous intratympanic dexamethasone delivered via a round window catheter for severe to profound sudden idiopathic sensorineural hearing loss after failure of systemic therapy. Laryngoscope. 2009 Feb;119(2):359-69. doi: 10.1002/lary.20074. PMID 19172627